## **Informed Consent Form**

| Protocol: SCRIPT | | | |
|---|---|---|---|
| Study Doctor: | | Site/Institution: Kings College London | |
| Participant Number: | | Participant Initials: | |
| Short Title: SRC inhibition as a potential target for Parkinson's disease psychosis | | | |
| By signing below you are confirming that you have read the participant information sheet and this informed consent form and understand it. | | | |
| I de | clare the following: | | |
| | | Please initial e | ach box. |
| • | | sheet dated <b>XXXX (version 1.0)</b> for the above e to ask questions about the study and my sfaction. | |
| • | • | cudy voluntarily and I can withdraw from the on, without penalty, losing any benefits and sing affected. | |
| • | • | vith additional contact details should I have or in the event of an illness that I think is | |
| • | | about me taking part in this study and they about my health, and that they may be fied during the study assessments. | |
| • | there be any concerns with what is four forwarded to the appropriate specialist for | n scan is not a diagnostic procedure. Should and however, I consent to my scans being or review and reporting. I further consent to to my General Practitioner and the research | |
| • | individuals from King's College London, fo | my medical notes may be looked at by rom regulatory authorities or from the NHS rt in this research. I give permission for these | |

I understand that my personal health information can be used and transferred in the

ways described previously.

| • | I specifically agree to my personal health information, collected during the study being sent outside the Euro described in this information sheet where laws don't prextent as the GDPR in the UK/EEA, but the Sponsor will protect my privacy. | pean Economic Ar<br>otect my privacy t | ea (EEA) as<br>to the same | |
|---|---|---|---|---|
| • | I understand that the information collected about me research in the future and shared anonymously with other | • | pport other | |
| • I understand that the Sponsor and other companies and people working for or with the Sponsor may use my personal health information in the future to: | | | | |
| 0 | study other therapies for patients; | | | |
| 0 | o develop a better understanding of diseases included in the study; and | | | |
| o | o improve the efficiency, design and methods of future clinical studies. | | | |
| I understand that I will not lose any of my legal rights by signing this informed consent form. | | | | |
| • | I will receive a fully signed and dated copy of this inform | ned consent form. | | |
| • | I agree to take part in this study. | | | |
| Each | person signing this informed consent form must person | ally date their own | signature. | |
| By si | gning below, I agree that I would like to take part in the s | study. | | |
| <br>Nam | e of participant (print) | | | |
| Sign | ature of participant | | Date | - |
| Print | ted name of person obtaining informed consent | - | | |
| Sign | ature of person obtaining informed consent | Date | | |

When completed, 1 signed and dated original for participant; 1 signed and dated original for researcher site file; 1 signed and dated copy to be kept in medical notes.